CLINICAL TRIAL: NCT06027021
Title: Assessment of Hypoxia Before Radioembolization Treatment With 18F-FMISO PET
Acronym: ARTE-MISO
Status: Completed | Type: Observational
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Cigdem Soydal, Asc Prof, Ankara University
Other Study IDs: ARTE-MISO
Record Dates: First submitted 2023-08-31; First posted 2023-09-07 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Radioembolization; Radiotherapy; Cancer; Positron Emission Tomography
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Treatment group: Patients received radioembolization with hepatocellular cancer or colorectal cancer liver metastases
  Interventions: Diagnostic Test: 18F-Fluoromisonidazole PET

INTERVENTIONS:
Diagnostic Test: 18F-Fluoromisonidazole PET — Imaging of hypoxia before radioembolization with 18F-Fluoromisonidazole PET.

SUMMARY:
Hypoxia is a known factor for resistance to radiotherapy in tumors. Response to transarterial radioembolization is known to be variable between different patients even if the same dose of radiation was delivered. In this study the investigators aim to quantify the hypoxia in the primary and secondary tumors of liver with 18F-FMISO PET before radioembolization and to prove any effect of the hypoxia, if present, on the dose that should be delivered to tumor to ensure treatment response.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with colorectal carcinoma with liver metastasis or hepatocellular carcinoma.
* Is not eligible for surgery
* Above 18 years old
* The patients who are referred for transarterial radioembolization treatment to Ankara University School of Medicine Department of Nuclear Medicine.

Exclusion Criteria:

* Patients with ECOG performance score >1
* Claustrophobia
* Life expectancy shorter than 3 months
* Pregnant or breast-feeding patients

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The patients with hepatocellular carcinoma or colorectal carcinoma with liver metastasis who are referred for transarterial radioembolization to Ankara University School of Medicine Department of Nuclear Medicine will be enrolled for the trial.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2023-08-15 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-07-15 (Actual)

PRIMARY OUTCOMES:
Demonstrate the effect of the hypoxia in the success of the radioembolization treatment | 08/2024
  Demonstrate the effect of the hypoxia in the success of the radioembolization treatment
The effect of the hypoxia on the dose-response relationships and required doses to achieve treatment response in the hypoxic and non-hypoxic group. | 08/2024
  The effect of the hypoxia on the dose-response relationships and required doses to achieve treatment response in the hypoxic and non-hypoxic group.

CONTACTS AND LOCATIONS:
Overall Officials: Cigdem Soydal, MD, Principal Investigator — Ankara University
Locations (1):
- Ankara University, Ankara, Turkey (Türkiye)